CLINICAL TRIAL: NCT00845260
Title: Internet- Versus Group-Administered Cognitive Behavior Therapy for Panic Disorder in a Psychiatric Setting: A Randomized Equivalence Trial
Brief Title: Internet-Versus Group-Administered Cognitive Behavior Therapy for Panic Disorder
Acronym: IP2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Nils Lindefors, MD, PHD, professor, Karolinska Institutet, Stockholm County Council
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IP2; Dnr 04-034/4
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Panic Disorder
MeSH Terms: conditions — Panic Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Internet CBT (Experimental): Internet-based cognitive behavior therapy (CBT).
  Interventions: Behavioral: Internet-based cognitive behavior therapy (CBT).
- Group CBT (Experimental): Group cognitive behavior therapy (CBT).
  Interventions: Behavioral: Group CBT

INTERVENTIONS:
Behavioral: Internet-based cognitive behavior therapy (CBT). — Self-help program and guidance by psychologist via e-mail during 10 weeks.
  Arms: Internet CBT
Behavioral: Group CBT — Group cognitive behavior therapy (CBT) during 10 weeks.
  Arms: Group CBT

SUMMARY:
Panic Disorder with or without agoraphobia (PD/A) is a common, and unless it is treated, often chronic psychiatric disorder. The are effective pharmacological as well as psychological treatments for PD/A. Because of the lack of availability of the most effective psychological treatment, cognitive behavior therapy (CBT), self-help based CBT treatments have been developed. One of those are Internet-based CBT. The aim of this study is to compare the effectiveness of Internet and group CBT for PD/A in a regular psychiatric setting. 113 patients are consecutively and randomly assigned to either treatment (both lasting 10 weeks). The main outcome measure is the Panic Disorder Severity Scale(PDSS). The study hypothesis is that treatments will show equal effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Primary Panic Disorder with or without Agoraphobia (PD/A)

Exclusion Criteria:

* active substance abuse
* physiological etiology of panic symptoms
* under 18 years of age
* severe depression or suicidal ideation.
* if on drugs for PD, not having had a constant dosage for 2 months
* undergoing other cognitive behavioral treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2004-12; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Panic Disorder Severity Scale (PDSS) | Pre, post at 6-month follow-up

SECONDARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) Anxiety Sensitivity Index (ASI) Sheehan Disability Scale (SDS) | Pre, post and 6-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Nils Lindefors, MD, PhD, professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Department of Clinical Neuroscience, Section of psychiatry, Karolinska Hospital Solna R5, Stockholm, Sweden

REFERENCES:
- [Derived] Lonsdorf TB, Ruck C, Bergstrom J, Andersson G, Ohman A, Lindefors N, Schalling M. The COMTval158met polymorphism is associated with symptom relief during exposure-based cognitive-behavioral treatment in panic disorder. BMC Psychiatry. 2010 Nov 26;10:99. doi: 10.1186/1471-244X-10-99. PMID 21110842
- [Derived] Bergstrom J, Andersson G, Ljotsson B, Ruck C, Andreewitch S, Karlsson A, Carlbring P, Andersson E, Lindefors N. Internet-versus group-administered cognitive behaviour therapy for panic disorder in a psychiatric setting: a randomised trial. BMC Psychiatry. 2010 Jul 2;10:54. doi: 10.1186/1471-244X-10-54. PMID 20598127